CLINICAL TRIAL: NCT04797637
Title: Post-operative Patient Positioning Device for Improvement of Post-Operative Pain in Parturients Undergoing Cesarean Delivery: A Randomized Controlled Trial
Brief Title: Post-operative Patient Positioning Device for Improvement of Post-Operative Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: GSquared Medical, LLC (Industry)
Responsible Party: Principal Investigator, Lisa C. Zuckerwise, MD, Assistant Professor of Obstetrics and Gynecology, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 210266
Record Dates: First submitted 2021-03-09; First posted 2021-03-15 (Actual); Results first posted 2023-01-06 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Pain, Postoperative
Keywords: cesarean; c-section; postoperative pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Participants will be randomized in a 1:1 ratio using permutated blocks of 6. REDCap will be used for randomization, using an uploaded randomization sequence. A member of the study team will access REDCap to complete randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Treatment Group (Experimental): Patients randomized to the treatment group will have the ABBy device applied by study personnel at the time of randomization, followed by a continuation of usual postoperative care.
  Interventions: Device: ABBy® Adjustable Panniculus Retractor for Wound Care
- Standard of Care (No Intervention): The control group will have postoperative care per usual care

INTERVENTIONS:
Device: ABBy® Adjustable Panniculus Retractor for Wound Care — The ABBy (G-Squared Medical, Brentwood, TN) is an extended-wear panniculus retractor/tissue stabilizer that is intended for use postoperatively after abdominal procedure. It is placed directly onto patient skin, superior to a transverse incision, and is then used to elevate redundant tissues away from an incision or wound (https://www.gsquaredmedical.com/How-it-Works.html). The ABBy can be removed and replaced by patients and can be used for up to 10 days. This study aims to assess the effect of ABBy use on postoperative pain, pain medication requirement, and patient satisfaction, when used as a patient-positioning device in women following cesarean delivery.
  Other Names: Abby device
  Arms: Treatment Group

SUMMARY:
This paucity of evidence supporting or dissuading the use of postoperative abdominal support following cesarean section for the reduction of postoperative pain leaves important clinical questions unanswered. Additionally, there is an absence of long-term outcomes associated with the use of abdominal support devices. There remains a need for the development and implementation of nonpharmacologic methods for analgesia for women following cesarean sections, along with evidence-based recommendations regarding their use in postoperative patients. The ABBy (G-Squared Medical, Brentwood, TN) is an extended-wear panniculus retractor/tissue stabilizer that is intended for use postoperatively after abdominal procedure.

It is placed directly onto patient skin, superior to a transverse incision, and is then used to elevate redundant tissues away from an incision or wound (https://www.gsquaredmedical.com/How-it-Works.html). The ABBy can be removed and replaced by patients and can be used for up to 10 days. This study aims to assess the effect of ABBy use on postoperative pain, pain medication requirement, and patient satisfaction, when used as a patient-positioning device in women following cesarean delivery.

DETAILED DESCRIPTION:
BACKGROUND:

Postoperative pain has significant short- and long-term implications for parturients undergoing cesarean delivery. Poorly controlled postoperative pain can interfere with the women's ability to care for herself and her newborn in the immediate postoperative period, and can contribute to longer length of hospitalizations. Untreated pain is associated with persistent pain, postpartum depression, and greater opioid use.

It is well established that an individualized, multimodal analgesic plan for the management of postoperative pain following cesarean delivery is associated with superior pain relief and decreased opioid consumption. While different institutional guidelines influence general practice patterns, a combination of several medications acting on different receptors has been shown to be effective in decreasing postoperative pain. In 2018, the cesarean section rate in the United States was 31.9%, compared to 20.7% in 1996. As the cesarean delivery rate increases, it is becoming more pertinent to develop and incorporate nonpharmacologic practices for postoperative pain.

The use of abdominal binders as an adjunct to pharmacologic therapy for the management of postoperative pain following major abdominal surgery has previously been discussed in surgical literature.

The utility of abdominal support within the Obstetrics literature is both sparse and conflicting.

This paucity of evidence supporting or dissuading the use of postoperative abdominal support following cesarean section for the reduction of postoperative pain leaves important clinical questions unanswered. Additionally, there is an absence of long-term outcomes associated with the use of abdominal support devices. There remains a need for the development and implementation of nonpharmacologic methods for analgesia for women following cesarean sections, along with evidence-based recommendations regarding their use in postoperative patients. The ABBy (G-Squared Medical, Brentwood, TN) is an extended-wear panniculus retractor/tissue stabilizer that is intended for use postoperatively after abdominal procedure. It is placed directly onto patient skin, superior to a transverse incision, and is then used to elevate redundant tissues away from an incision or wound (https://www.gsquaredmedical.com/How-it-Works.html). The ABBy can be removed and replaced by patients and can be used for up to 10 days. This study aims to assess the effect of ABBy use on postoperative pain, pain medication requirement, and patient satisfaction, when used as a patient-positioning device in women following cesarean delivery.

ENROLLMENT/RANDOMIZATION:

All residents and Labor and Delivery staff will be apprised of the study and appropriate patients with either planned cesarean delivery or those delivered by cesarean delivery within 36 hours will have the opportunity to participate in the trial. The research team will use a daily list of all cesarean deliveries in Epic to identify potentially eligible patients for enrollment. Prior to contacting the patient, the research team member will check with the patient's nurse or care team to discuss eligibility and appropriateness for the study. Notices will also be placed in Labor and Delivery regarding the study. Study personnel will explain the study to the patient and allow ample time for the subject to ask questions related to the study. If the subject consents, she will sign the informed consent document and will be provided with a copy of the consent form prior to randomization.

Patients will be enrolled either during their delivery admission up until 36 hours after delivery. After enrolling, randomization will be performed on the obstetric unit within the first 36 hours postpartum. Participants will be randomized in a 1:1 ratio using permutated blocks of 6. REDCap will be used for randomization, using an uploaded randomization sequence. A member of the study team will access REDCap to complete randomization. The randomization result will be notated with the patient's study number and retained in the research record.

STUDY PROCEDURES:

Patients who meet inclusion criteria and undergo cesarean delivery at Vanderbilt University Hospital center will be asked to participate. Informed consent will be obtained during the delivery admission. Enrolled patients will be randomized within the first 36 hours following cesarean delivery. The 36-hour window for randomization will begin at the completion of surgical case, as marked in the Anesthetic Care Record in the EMR.

Patients randomized to the treatment group will have the ABBy device applied by study personnel at the time of randomization, followed by continuation of usual postoperative care. The control group will have postoperative care per usual care.

Cesarean delivery will be performed by patients' surgical team, with surgical technique per surgeon preference. Women in the treatment group will have the ABBy device placed above the incision within 36 hours of cesarean delivery completion. All team members placing the ABBy device will undergo training and demonstrate competence.

Postoperative analgesia will be administered to all participants as per routine guidelines on postpartum. All study patients will receive an electronic survey at 10 days postoperatively and again at 14 days for those continuing to use the ABBy device or opioid medication at the 10-day survey.

Specific medical information regarding pregnancy and delivery will be collected and analyzed from the patients' electronic medical records.

RISKS:

A rare risk exists if the patient has an unknown allergy to the adhesive material in the device, though this is estimated at less than one per one million for the silicone-based adhesive used, and per the manufacturer's report, the raw materials used in the silicone roll stock construction (PS-1860) have been analyzed for biocompatibility and found to not cause any adverse effect when used properly (Polymer Science, Monticello, IN).

There is a risk of confidentiality breech in the collection of medical information. All efforts will be made to protect the personal information of the patient by the use of study number assignment and a password-protected database. Any breech in confidentiality will be promptly reported to the Vanderbilt IRB.

Any adverse events will be reported to the Institutional Review Board in a timely manner as appropriate.

STUDY WITHDRAWAL/DISCONTINUATION:

Any patient who wishes to withdraw from the study will be allowed to withdraw. Should the patient decide to withdraw from the study, she will notify the principal investigator and her information will be deleted from the study records.

STATISTICAL CONSIDERATIONS:

Sample size: To detect a reduction in pain medication use of 40% using an alpha of 0.05 and a beta of 0.20, 108 patients per group with a total sample of 216 patients will be required. The labor and delivery unit performs about 1400 cesarean deliveries annually; therefore, assuming an 80% eligibility rate and subsequent 50% participation rate, the study would be conducted over a 12-month period.

PRIVACY/CONFIDENTIALITY:

Risks to participants are minimized by limiting this prospective study to subjects meeting the inclusion/exclusion criteria. Access to PHI will be limited to the PI and co-investigators. All patients will be de-identified by assignment of a study number. All data collected in this study will be kept electronically in a secure REDCap database. The primary risk in this study involves the disclosure of protected health information. This risk is reasonable, given the above precautions, in relation to the potential benefit to both future patients and society in general by the possibility of reducing the use of pain medication in cesarean patients.

FOLLOW-UP/RECORD RETENTION:

The study will require 1 year for complete enrollment. Participants will be actively enrolled in the study for the duration of their or delivery admission plus up to 14 days follow-up time. Research records will be retained for up to 6 years.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years
2. Cesarean delivery
3. <36 hours post-delivery

Exclusion Criteria:

1. Vertical skin incision
2. Inability to place device superior to incision
3. Presence of surgical drain
4. Opioid use disorder
5. Chronic opioid use (> 14 consecutive days during pregnancy)
6. Allergy to device adhesive
7. Active COVID-19 infection
8. Patient unable to consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — This is a obstetric study and only affects women.
Enrollment: 278 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-07-20 (Actual); Study Completion 2022-07-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Zuckerwise, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] ACOG Committee Opinion No. 742: Postpartum Pain Management. Obstet Gynecol. 2018 Jul;132(1):e35-e43. doi: 10.1097/AOG.0000000000002683. PMID 29781876
- [Background] Corso E, Hind D, Beever D, Fuller G, Wilson MJ, Wrench IJ, Chambers D. Enhanced recovery after elective caesarean: a rapid review of clinical protocols, and an umbrella review of systematic reviews. BMC Pregnancy Childbirth. 2017 Mar 20;17(1):91. doi: 10.1186/s12884-017-1265-0. PMID 28320342
- [Background] Eisenach JC, Pan PH, Smiley R, Lavand'homme P, Landau R, Houle TT. Severity of acute pain after childbirth, but not type of delivery, predicts persistent pain and postpartum depression. Pain. 2008 Nov 15;140(1):87-94. doi: 10.1016/j.pain.2008.07.011. Epub 2008 Sep 24. PMID 18818022
- [Background] Chou R, Gordon DB, de Leon-Casasola OA, Rosenberg JM, Bickler S, Brennan T, Carter T, Cassidy CL, Chittenden EH, Degenhardt E, Griffith S, Manworren R, McCarberg B, Montgomery R, Murphy J, Perkal MF, Suresh S, Sluka K, Strassels S, Thirlby R, Viscusi E, Walco GA, Warner L, Weisman SJ, Wu CL. Management of Postoperative Pain: A Clinical Practice Guideline From the American Pain Society, the American Society of Regional Anesthesia and Pain Medicine, and the American Society of Anesthesiologists' Committee on Regional Anesthesia, Executive Committee, and Administrative Council. J Pain. 2016 Feb;17(2):131-57. doi: 10.1016/j.jpain.2015.12.008. PMID 26827847
- [Background] Martin JA, Hamilton BE, Osterman MJK, Driscoll AK. Births: Final Data for 2018. Natl Vital Stat Rep. 2019 Nov;68(13):1-47. PMID 32501202
- [Background] Stoker KC. Use of Abdominal Binders for Postoperative Pain After Gastrointestinal Surgery: An Integrative Review. J Perianesth Nurs. 2019 Aug;34(4):829-833. doi: 10.1016/j.jopan.2018.10.010. Epub 2019 Feb 7. PMID 30745077
- [Background] Ossola P, Mascioli F, Coletta D, Pizzato M, Bononi M. Evidence on postoperative abdominal binding: A systematic review with meta-analysis of randomized controlled trials. Surgeon. 2021 Aug;19(4):244-251. doi: 10.1016/j.surge.2020.07.003. Epub 2020 Aug 6. PMID 32773235
- [Background] Gillier CM, Sparks JR, Kriner R, Anasti JN. A randomized controlled trial of abdominal binders for the management of postoperative pain and distress after cesarean delivery. Int J Gynaecol Obstet. 2016 May;133(2):188-91. doi: 10.1016/j.ijgo.2015.08.026. Epub 2016 Jan 14. PMID 26892694
- [Background] Gustafson JL, Dong F, Duong J, Kuhlmann ZC. Elastic Abdominal Binders Reduce Cesarean Pain Postoperatively: A Randomized Controlled Pilot Trial. Kans J Med. 2018 May 18;11(2):1-19. eCollection 2018 May. PMID 29796155
- [Derived] Zuckerwise LC, Mulhall JC, Thompson JL, Jackson LA, McNeill-Simaan EO, Osmundson SS. Effect of panniculus elevation device on postoperative pain after cesarean delivery: a randomized controlled trial. Am J Obstet Gynecol MFM. 2023 May;5(5):100920. doi: 10.1016/j.ajogmf.2023.100920. Epub 2023 Mar 6. PMID 36889439

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients who meet inclusion criteria and undergo cesarean delivery at Vanderbilt University Hospital center will be asked to participate. Informed consent will be obtained during the delivery admission. Enrolled patients will be randomized within the first 36 hours following cesarean delivery. Recruitment will occur from 4/1/2020-7/31/2021 or until enrollment target achieve.
Period: Overall Study
Arm/Group | Treatment Group | Standard of Care
Started | 141 | 137
Completed | 118 | 104
Not Completed | 23 | 33
Not completed — Lost to Follow-up | 23 | 32
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Group | Standard of Care | Total
Number analyzed (Participants) | 118 | 104 | 222
Age, Continuous [Median (Inter-Quartile Range); unit: Years] | 31 [27 to 36] | 31 [26 to 34] | 31 [26 to 35]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 118 | 104 | 222
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 75 | 67 | 142
  Black | 20 | 14 | 34
  Hispanic | 8 | 7 | 15
  Asian | 3 | 6 | 9
  Multiracial or unknown | 12 | 10 | 22
Parity [Median (Inter-Quartile Range); unit: Pregnancies] | 2 [1 to 2] | 1 [1 to 2] | 2 [1 to 2]
BMI at delivery [Median (Inter-Quartile Range); unit: Kg/M2] | 33 [29 to 37] | 34 [29 to 38] | 33 [29 to 44]
Completed high school education or less [Count of Participants; unit: Participants] | 34 | 36 | 70
Depression or anxiety [Count of Participants; unit: Participants] | 40 | 32 | 72
Tobacco use in pregnancy [Count of Participants; unit: Participants] | 7 | 3 | 10
Prior cesarean delivery [Count of Participants; unit: Participants] | 44 | 33 | 77

OUTCOME MEASURES:

1. Primary Outcome: Total Morphine Milliequivalent (MME) Use Postoperatively After Cesarean Delivery
Description: Postoperative analgesia will be administered to all participants as per routine guidelines on postpartum.
Time Frame: 14 days postoperative
Measure: Median (Inter-Quartile Range); unit: Morphine milligram equivalents
Arm/Group | Treatment Group | Standard of Care
Number analyzed (Participants) | 118 | 104
Morphine milligram equivalents | 52 [15 to 112] | 68 [18 to 112]

2. Secondary Outcome: Subjective Pain Scores During Use of Patient Positioning Device
Description: Postoperative analgesia will be administered to all participants as per routine guidelines on postpartum. All study patients will receive an electronic survey at 10 days postoperatively and again at 14 days for those continuing to use the ABBy device or opioid medication at the 10-day survey.
  Subjective pain scores (zero to 100 sliding scale) Please provide a number that best describes pain you have experienced at its WORST since discharge? No pain (0) worst pain imaginable (100) Please provide a number that best describes the AVERAGE pain you have experienced since discharge? No pain (0) worst pain imaginable (100)
Time Frame: Baseline to 14 days postoperative
Measure: Median (Inter-Quartile Range); unit: score on a scale (0-100)
Arm/Group | Treatment Group | Standard of Care
Number analyzed (Participants) | 118 | 104
score on a scale (0-100)
  Pain at worst | 50 [27 to 66] | 51 [20 to 73]
  Average pain experienced | 25 [15 to 35] | 30 [11 to 50]

3. Secondary Outcome: Patient Satisfaction During Use of Patient Positioning Device.
Description: Postoperative analgesia will be administered to all participants as per routine guidelines on postpartum. All study patients will receive an electronic survey at 10 days postoperatively and again at 14 days for those continuing to use the ABBy device or opioid medication at the 10-day survey.
  Patient satisfaction with device
  Question as part of a survey to patients who had the ABBy device placed:
  I would use ABBy next time (strongly agree, agree, neutral, disagree, strongly disagree)
Time Frame: Baseline to 14 days postoperative
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group
Number analyzed (Participants) | 100
Participants
  Strongly agree | 30
  Agree | 33
  Neutral | 24
  Disagree | 12
  Strongly disagree | 1

4. Secondary Outcome: Duration of Use of Patient Positioning Device.
Description: Postoperative analgesia will be administered to all participants as per routine guidelines on postpartum. All study patients will receive an electronic survey at 10 days postoperatively and again at 14 days for those continuing to use the ABBy device or opioid medication at the 10-day survey.
  Duration of use of patient positioning device Question on survey: How long did you use the ABBy? (please enter a number of days, counting from the day placed as zero)
Time Frame: Baseline to 14 days postoperative
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Treatment Group
Number analyzed (Participants) | 63
Days | 5 [3 to 9]

5. Secondary Outcome: Number of Participants With Surgical Complications in Groups With and Without Patient Positioning Device
Description: Specific medical information regarding pregnancy and delivery will be collected and analyzed from the patients' electronic medical records.
Time Frame: Baseline to 14 days
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group | Standard of Care
Number analyzed (Participants) | 118 | 104
Participants
  endometritis | 1 | 1
  Problems with the incision healing | 2 | 0
  mastitis | 0 | 0
  venous thromboembolism | 0 | 0
  postpartum hemorrhage | 0 | 0
  6. Postpartum preeclampsia | 3 | 2

6. Secondary Outcome: Surgical Costs in Groups With and Without Patient Positioning Device
Description: Additional costs resulting from surgical complications.
Time Frame: Baseline to 14 days
Population: Due to the inability to achieve the necessary sample size of surgical complications, there was no data collected to analyze the costs.
Arm/Group | Treatment Group | Standard of Care
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 14 days
Arm/Group | Treatment Group | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/118 | 0/104
Serious Adverse Events (participants affected / at risk) | 0/118 | 0/104
Other Adverse Events (participants affected / at risk) | 10/118 | 6/104
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Group (N=118) | Standard of Care (N=104)
Since, discharge have you had any complications related to your delivery? (Surgical and medical procedures) | 10 (10) | 6 (6) — Yes/No, If yes, what were those complications? Infection of the uterus Breast infection Blood clot Excessive bleeding
Problems with the incision (Surgical and medical procedures) | 2 (2) | 0 (0)
Infection of the uterus (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 2 (2)
Breast infection (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0)
Blood clot (Blood and lymphatic system disorders) | 0 (0) | 0 (0)
Excessive bleeding (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0)
Other (Pregnancy, puerperium and perinatal conditions) | 8 (8) | 4 (4) — preeclampsia, postpartum depression/anxiety, anesthesia complications (nerve injury, postdural puncture headache)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-16): https://cdn.clinicaltrials.gov/large-docs/37/NCT04797637/Prot_SAP_000.pdf